CLINICAL TRIAL: NCT03111498
Title: Technical Skills Training Programme for Conducting Vacuum Assisted Deliveries - a Randomized Controlled Trial
Brief Title: Technical Skills Training Programme for Conducting Vacuum Assisted Deliveries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich Husslein (Other)
Responsible Party: Sponsor-Investigator, Heinrich Husslein, Ass-Prof., MD, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2300/2016
Record Dates: First submitted 2017-03-15; First posted 2017-04-12 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Training VAD
Keywords: Vacuum assisted delivery; technical skills; training

STUDY DESIGN:
Intervention Model Description: video-recorded vacuum procedure on a special VAD-training phantom in a randomized setting: (1) theory-based training programme (2) practice-based training programme (one-to-one teaching).
  Video-recorded vacuum procedure on the VAD- training phantom before randomization, directly after training programme, 4-8 weeks after training programme in order to determine retention of skills.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- theory-based training programme (Other): theory-based training programme (oral presentation including a step-by-step guidance saying)
  Interventions: Other: theory-based training programme
- practice-based training (Other): practice-based training programme (one-to-one teaching)
  Interventions: Other: practice-based training programme (one-to-one teaching)

INTERVENTIONS:
Other: practice-based training programme (one-to-one teaching) — practice-based training programme (one-to-one teaching) for conducting VAD
  Arms: practice-based training
Other: theory-based training programme — theory-based training programme for conducting VAD
  Arms: theory-based training programme

SUMMARY:
Training is very important for acquisition and maintenance of obstetric skills. As a one-to-one practical teaching needs time and personal resources, the investigators want to prove the benefit and necessity of the one-to-one training program compared to a theory-based training program in conducting vacuum assisted deliveries (VAD).

The aim of this study is to prove that a practice-based training program (one-to- one teaching) leads to better training results compared to a theory-based training program in conducting VAD.

ELIGIBILITY:
Inclusion Criteria:

* employees of the Department of Obstetrics and Gynaecology
* oral and written informed consent

Exclusion Criteria:

* no oral and written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
technical skills in conducting VAD | one day (day 0)
  General and procedure-specific skills will be assessed using a validated rating tool.

SECONDARY OUTCOMES:
Retention of skills conducting VAD | 4-8 weeks after day 0
  General and procedure-specific skills will be assessed using a validated rating tool.
trainees' satisfaction | 4-8 weeks after day 0
  trainees' satisfaction with the two different training programmes will be assessed using a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Julian Marschalek, MD, Study Chair — Medical University of Vienna
Locations (1):
- Dept. Obstetrics and Gynaecology, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided